CLINICAL TRIAL: NCT04791319
Title: A Phase 2b, Multicenter, Randomized, Placebo- and Active-comparator-controlled, Double-blind Study to Evaluate the Safety and Efficacy of Bermekimab (JNJ-77474462) for the Treatment of Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Bermekimab (JNJ-77474462) in the Treatment of Participants With Moderate to Severe Atopic Dermatitis
Acronym: GENESIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature Termination due to Interim Analysis (100 patients at Week 16) meeting futility.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108932; 2020-002587-31 (EudraCT Number); 77474462ADM2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-03-09; First posted 2021-03-10 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — bermekimab; dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Placebo (Placebo Comparator): Participants will receive subcutaneous (SC) placebo once a week (qw) through Week 15. At Week 16, participants will crossover to receive SC bermekimab Dose 2 qw through Week 31.
  Interventions: Drug: Placebo; Drug: Bermekimab
- Group 2: Bermekimab (Experimental): Participant will receive SC bermekimab Dose 1 qw from Week 0 through Week 31.
  Interventions: Drug: Bermekimab
- Group 3: Bermekimab (Experimental): Participants will receive SC bermekimab Dose 2 qw from Week 0 through Week 15. At Week 16, participants who achieve an eczema area and severity index (EASI)-75 response (responders) will be rerandomized either to continue to receive bermekimab Dose 2 qw, or to receive bermekimab Dose 1 qw, through Week 31 and participants who do not achieve an EASI-75 response (non responders) will continue to receive bermekimab Dose 2 qw through Week 31.
  Interventions: Drug: Bermekimab
- Group 4: Dupilumab (Active Comparator): Participants will receive a loading dose of SC dupilumab Dose 1 at Week 0, SC placebo every two week (q2w) from Week 1 through Week 15 and then dupilumab Dose 2 q2w from Week 2 through Week 14. At Week 16, participants who achieve EASI-75 response (dupilumab responders) will continue on dupilumab Dose 2 q2w through Week 30 and placebo q2w from Week 17 through Week 31. Participants who do not achieve an EASI-75 response (dupilumab non-responders) will receive placebo qw from Week 16 through Week 18 (washout period) and bermekimab Dose 2 qw from Week 19 through Week 31.
  Interventions: Drug: Placebo; Drug: Bermekimab; Drug: Dupilumab

INTERVENTIONS:
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Group 1: Placebo; Group 4: Dupilumab
Drug: Bermekimab — Bermekimab will be administered subcutaneously.
  Other Names: JNJ-77474462
Drug: Dupilumab — Dupilumab will be administered subcutaneously.
  Arms: Group 4: Dupilumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of bermekimab in participants with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Be otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiograms (ECGs) performed at screening. Any abnormalities, must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Have atopic dermatitis (AD) for at least 1 year (365 days) prior to the first administration of study intervention as determined by the investigator through participant interview and/or review of the medical history
* Have a history of inadequate response to treatment for AD with topical medications or for whom topical treatments are otherwise medically inadvisable (example [eg], due to important side effects or safety risks)
* Be considered, in the opinion of the investigator, a suitable candidate for dupilumab (DUPIXENT) therapy according to their country's approved DUPIXENT product labeling
* Have an eczema area and severity index (EASI) score greater than or equal (>=) to 16 at screening and at baseline
* Have an investigator global assessment (IGA) score >=3 and involved body surface area (BSA) >=10 percent (%) at screening and baseline

Exclusion Criteria:

* Has a current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has unstable cardiovascular disease, defined as a recent clinical deterioration (eg, unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months
* Has or has had a serious infection (eg, sepsis, pneumonia, or pyelonephritis), or has been hospitalized or received intravenous (IV) antibiotics for an infection during the 2 months before screening
* Has or has had herpes zoster within the 2 months before screening
* Has a history of being human immunodeficiency virus (HIV) antibody-positive, or tests positive for HIV at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (42):
- United States (18):
  - California Allergy & Asthma Medical Group Inc., Los Angeles, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Park Avenue Dermatology, Orange Park, Florida
  - Forcare Clinical Research, Inc., Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Grekin Skin Institute, Warren, Michigan
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island
  - Arlington Center for Dermatology, Arlington, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Clinical Research, Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
- Canada (6):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Allergy Research Canada Inc., Niagara Falls, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre De Recherche Dermatologique Du Quebec Metropolitan, Québec, Quebec
- Germany (8):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Goethe Universität Frankfurt, Frankfurt am Main
  - TFS Trial Form Support GmbH, Hamburg
  - MensingDerma research GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Praxis Dr. med. Beate Schwarz - Germany, Langenau
  - Hautarztpraxis, Mahlow
- Japan (3):
  - Takagi Clinic, Obihiro-shi
  - Kume Clinic, Osaka Fu
  - Sapporo Skin Clinic, Sapporo
- Poland (7):
  - Nzoz Przychodnia Specjalistyczna Medica, Częstochowa
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - DermoDent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski s.c., Osielsko
  - Klinika Ambroziak Estederm Sp. z o.o, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Centrum Medyczne Matusiak w CITYCLINICPrzychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw
  - WroMedica I.Bielicka, A.Strzałkowska s.c., Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received two placebo subcutaneous (SC) injections once a week (qw) from Week 0 through Week 15.
- Bermekimab 350 mg: Participants received a single bermekimab 350 milligrams (mg) SC injection qw from Week 0 through Week 15.
- Bermekimab 700 mg: Participants received bermekimab 700 mg (2 doses of 350mg) SC injections qw from Week 0 through Week 15.
- Dupilumab: Participants received a loading dose of dupilumab 600 mg (2 doses of 300 mg) SC injection at Week 0 followed by two placebo SC injections every two weeks (q2w) from Week 1 through Week 15 and a single dupilumab 300 mg SC injection q2w beginning at Week 2 through Week 14.
- Placebo Then Bermekimab 700 mg: After completion of placebo-contorlled period, at Week 16 participants entered active treatment period and were crossed-over to receive bermekimab 700 mg (2 doses of 350 mg) SC injection qw through Week 31.
- Bermekimab 350 mg Then Bermekimab 350 mg: After completion of placebo-controlled period, at Week 16 participants entered active treatment period and continued to receive a single bermekimab 350 mg SC injection qw through 31.
- Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders): After completion of placebo-controlled period, at Week 16 participants who did not achieved an eczema area and severity index (EASI-75) response (greater than or equal to [>=] 75 percent [%] improvement from baseline) were considered as non-responders and they continued bermekimab 700 mg SC injection qw through Week 31.
- Bermekimab 700 mg Then Bermekimab 700 mg (Responders): After completion of placebo-controlled period, at Week 16 participants who achieved an EASI-75 response were considered as responders and were rerandomized to receive bermekimab 700 mg (2 doses of 350 mg) SC injection qw through Week 31.
- Bermekimab 700 mg Then Bermekimab 350 mg (Responders): After completion of placebo-controlled period, at Week 16 participants who achieved an EASI-75 response were considered as responders and were rerandomized to receive bermekimab 350 mg SC injection qw through Week 31.
- Dupilumab Then Dupilumab 300 mg (Responders): After completion of placebo-controlled period, at Week 16 participants who achieved an EASI-75 response were considered as responders and they continued to dupilumab 300 mg SC injection q2w from Week 16 through Week 30 and placebo SC injection q2w from Week 17 through Week 31.
- Dupilumab Then Bermekimab 700 mg (Non-Responders): After completion of placebo-controlled period, at Week 16 participants who did not achieved an EASI-75 response were considered as non-responders and they received placebo SC injection qw from Week 16 through Week 18 (that is, washout period), and bermekimab 700 mg SC injection qw from Week 19 through Week 31.
Period: Placebo Controlled Period (Week 0-15)
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab | Placebo Then Bermekimab 700 mg | Bermekimab 350 mg Then Bermekimab 350 mg | Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) | Dupilumab Then Dupilumab 300 mg (Responders) | Dupilumab Then Bermekimab 700 mg (Non-Responders)
Started | 33 | 33 | 67 | 66 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 33 | 33 | 67 | 65 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 19 | 21 | 30 | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 12 | 37 | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Trial termination | 2 | 4 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participants who completed only safety follow-up | 7 | 6 | 21 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Period (Week 16-31)
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab | Placebo Then Bermekimab 700 mg | Bermekimab 350 mg Then Bermekimab 350 mg | Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) | Dupilumab Then Dupilumab 300 mg (Responders) | Dupilumab Then Bermekimab 700 mg (Non-Responders)
Started | 0 | 0 | 0 | 0 | 19 | 21 | 22 | 3 | 5 | 27 | 11
Completed | 0 | 0 | 0 | 0 | 1 | 6 | 3 | 1 | 1 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 18 | 15 | 19 | 2 | 4 | 21 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Trial termination and COVID-19 related | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 0 | 1 | 9 | 2
Not completed — Participants who completed safety follow-up | 0 | 0 | 0 | 0 | 12 | 8 | 16 | 2 | 3 | 11 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized at Week 0 and received at least 1 dose of study intervention.
Groups:
- Placebo: Participants received two placebo subcutaneous (SC) injections once a week (qw) through Week 15. After completion of placebo-contorlled period, at Week 16 participants entered active treatment period and were crossed-over to receive bermekimab 700 mg (2 doses of 350 mg) SC injection qw through Week 31.
- Bermekimab 350 mg: Participants received a single bermekimab 350 milligrams (mg) SC injection qw from Week 0 through Week 15. After completion of placebo-controlled period, at Week 16 participants entered active treatment period and continued to receive a single bermekimab 350 mg SC injection qw through 31.
- Bermekimab 700 mg: Participants received bermekimab 700 mg (2 doses of 350mg) SC injections qw from Week 0 through Week 15. After completion of placebo-controlled period, at Week 16 participants who achieved an eczema area and severity index (EASI-75) response (greater than or equal to [>=] 75 percent [%] improvement from baseline) were considered as responders and were rerandomized in a 1:1 ratio either to receive bermekimab 700 mg (2 doses of 350 mg) SC injection qw or to receive bermekimab 350 mg SC injection qw through Week 31. After completion of placebo-controlled period, at Week 16 participants who did not achieved an EASI-75 response were considered as non-responders and they continued bermekimab 700 mg SC injection qw through Week 31.
- Dupilumab: Participants received a loading dose of dupilumab 600 mg (2 doses of 300 mg) SC injection at Week 0 followed by two placebo SC injections every two weeks (q2w) from Week 1 through Week 15 and a single dupilumab 300 mg SC injection q2w beginning at Week 2 through Week 14. After completion of placebo-controlled period, at Week 16 participants who achieved an EASI-75 response were considered as responders and they continued to dupilumab 300 mg SC injection q2w from Week 16 through Week 30 and placebo SC injection q2w from Week 17 through Week 31. After completion of placebo-controlled period, at Week 16 participants who did not achieved an EASI-75 response were considered as non-responders and they received placebo SC injection qw from Week 16 through Week 18 (that is, washout period), and bermekimab 700 mg SC injection qw from Week 19 through Week 31.
- Total: Total of all reporting groups
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab | Total
Number analyzed (Participants) | 33 | 33 | 67 | 65 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (14.18) | 34.6 (13.32) | 36 (12.3) | 37.2 (15.02) | 36 (13.65)
Age, Customized [Count of Participants; unit: Participants]
  From 18 to 64 years | 33 | 33 | 66 | 62 | 194
  From 65 to 84 years | 0 | 0 | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 28 | 32 | 87
  Male | 20 | 19 | 39 | 33 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 4 | 9
  Not Hispanic or Latino | 33 | 31 | 62 | 59 | 185
  Unknown or Not Reported | 0 | 2 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 7 | 14 | 10 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 2 | 7 | 12
  White | 25 | 20 | 51 | 46 | 142
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 2 | 0 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  CANADA | 8 | 6 | 15 | 15 | 44
  GERMANY | 8 | 8 | 14 | 14 | 44
  JAPAN | 2 | 4 | 7 | 4 | 17
  POLAND | 10 | 12 | 19 | 21 | 62
  UNITED STATES | 5 | 3 | 12 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index-75 (EASI-75) (Greater Than or Equal to [>=] 75 Percent [%] Improvement From Baseline) at Week 16
Description: Percentage of participants achieving EASI-75 at Week 16 were reported. EASI-75 response is defined as at least 75% improvement from baseline in EASI total score. The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Week 16
Population: The modified full analysis set (mFAS) included all participants who were randomized at Week 0 and received at least 1 dose of study intervention and had reached a visit by the time of the decision was made to terminate the study on 02 February 2022. Participants were excluded from the analysis after projected visit. Projected visit (weeks) = (decision date of study termination - first dose date +1) /7.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab
Number analyzed (Participants) | 21 | 24 | 42 | 43
percentage of participants | 9.5 | 16.7 | 16.7 | 51.2
Statistical Analysis 1: Comparison: Placebo vs Bermekimab 350 mg; Test type: Superiority; p = 0.489, Chi-squared — Threshold for significance at 0.05 level; MH weights = 7.1, 95% CI 2-sided [-12.1 to 26.2]
Statistical Analysis 2: Comparison: Placebo vs Bermekimab 700 mg; Test type: Superiority; p = 0.448, Chi-squared; MH Weights = 7.1, 95% CI 2-sided [-9.4 to 23.7]
Statistical Analysis 3: Comparison: Placebo vs Dupilumab; Test type: Superiority; p = 0.001, Chi-squared; MH Weights = 42.0, 95% CI 2-sided [22.9 to 61.1]

2. Secondary Outcome: Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 and a Reduction From Baseline of >=2 Points at Week 16
Description: Percentage of participants achieving vIGA-AD at Week 16 were reported. It is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0, where 0=Clear: No inflammatory signs of AD; 1=almost clear: Barely perceptible erythema, induration/papulation and/or lichenification; 2=mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting; 3=moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present and 4=severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present. Higher score indicated more severity of AD.
Time Frame: Week 16
Population: The mFAS included all participants who were randomized at Week 0 and received at least 1 dose of study intervention and had reached a visit by the time of the decision was made to terminate the study on 02 February 2022. Participants were excluded from the analysis after projected visit. Projected visit (weeks) = (decision date of study termination - first dose date +1) /7.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab
Number analyzed (Participants) | 21 | 24 | 42 | 43
percentage of participants | 9.5 | 12.5 | 11.9 | 27.9

3. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) in Eczema-Related Itch Numeric Rating Scale (NRS) of Score >=4 at Week 16 Among Participants With a Baseline Itch Value >=4
Description: Percentage of participants with improvement (reduction from baseline) in eczema-related itch NRS of score >=4 at Week 16 among participants with a baseline itch value >=4 were reported. The eczema skin pain and Itch NRS is a 2-item patient-reported outcome that participants used to rate the severity of their eczema-related skin pain and eczema related itch daily. Participants were asked the following questions: Please rate the severity of your eczema-related skin pain at its worst in the past 24 hours; and please rate the severity of your eczema-related itch at its worst in the past 24 hours. Each item was on a 0 to 10 NRS ranging from 0 "none" to 10 "worst possible" and were scored separately. Higher score indicated more severity.
Time Frame: Week 16
Population: The mFAS included all participants who were randomized at Week 0 and received at least 1 dose of study intervention and had reached a visit by the time of the decision was made to terminate the study on 02 February 2022. Participants were excluded from the analysis after projected visit. Projected visit (weeks) = (decision date of study termination - first dose date +1) /7. Here, N (number of participants analyzed) signifies participants who were evaluated for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab
Number analyzed (Participants) | 19 | 20 | 32 | 34
percentage of participants | 10.5 | 20.0 | 6.3 | 32.4

4. Secondary Outcome: Percentage of Participants Achieving EASI-90 (>= 90% Improvement in EASI From Baseline) at Week 16
Description: Percentage of participants achieving EASI-90 at Week 16 were reported. EASI-90 response is defined as at least 90% improvement from baseline in EASI total score. The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration/papulation, excoriation and lichenification on 4 anatomic regions of the body: head/neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab
Number analyzed (Participants) | 21 | 24 | 42 | 43
percentage of participants | 9.5 | 12.5 | 11.9 | 34.9

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were AEs with onset during the intervention period or that were a consequence of a pre-existing condition that has worsened since baseline. AEs are presented by individual dose received by participants during placebo-controlled period and by responders individual dose received during active treatment period.
Time Frame: Up to Week 36
Population: The safety analysis set included all participants who had received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Bermekimab 350 mg: Participants received a single bermekimab 350 milligrams (mg) SC injection qw from Week 0 through Week 15. After completion of placebo-controlled period, at Week 16 participants entered active treatment period and continued to receive a single bermekimab 350 mg SC injection qw through 31. Participants who received bermekimab 350 mg from Week 0 to Week 15 and continued to receive bermekimab 350 mg from Week 16 to Week 31 were combined in this arm.
- Bermekimab 700 mg: Participants received bermekimab 700 mg (2 doses of 350mg) SC injections qw from Week 0 through Week 15. After completion of placebo-controlled period, at Week 16 participants who did not achieved an eczema area and severity index (EASI-75) response (greater than or equal to [>=] 75 percent [%] improvement from baseline) were considered as non-responders and they continued bermekimab 700 mg SC injection qw through Week 31. After completion of placebo-controlled period, at Week 16 participants who achieved an EASI-75 response were considered as responders and were rerandomized to receive bermekimab 700 mg (2 doses of 350 mg) SC injection qw through Week 31. Participants who received bermekimab 700 mg from Week 0 to Week 15 and continued to receive bermekimab 700 mg from Week 16 to Week 36 (responders and non-responders) were combined in this arm.
- Dupilumab: Participants received a loading dose of dupilumab 600 mg (2 doses of 300 mg) SC injection at Week 0 followed by two placebo SC injections every two weeks (q2w) from Week 1 through Week 15 and a single dupilumab 300 mg SC injection q2w beginning at Week 2 through Week 14. After completion of placebo-controlled period, at Week 16 participants who achieved an EASI-75 response were considered as responders and they continued to dupilumab 300 mg SC injection q2w from Week 16 through Week 30 and placebo SC injection q2w from Week 17 through Week 31. Participants who received dupilumab 300 mg from Week 1 to Week 15 and continued to receive dupilumab 300 mg from Week 16 to Week 30 were combined in this arm.
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab | Placebo Then Bermekimab 700 mg | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) | Dupilumab Then Bermekimab 700 mg (Non-Responders)
Number analyzed (Participants) | 33 | 33 | 67 | 65 | 19 | 5 | 11
Participants | 18 | 26 | 46 | 40 | 7 | 2 | 4

6. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. Any SAE with onset during the intervention period or that were a consequence of a pre-existing condition that has worsened since baseline was considered to be TESAEs. AEs are presented by individual dose received by participants during placebo-controlled period and active treatment period.
Time Frame: Up to Week 36
Population: The safety analysis set included all participants who had received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab | Placebo Then Bermekimab 700 mg | Bermekimab 350 mg Then Bermekimab 350 mg | Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) | Dupilumab Then Dupilumab 300 mg (Responders) | Dupilumab Then Bermekimab 700 mg (Non-Responders)
Number analyzed (Participants) | 33 | 33 | 67 | 65 | 19 | 21 | 22 | 3 | 5 | 27 | 11
Participants | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Serum Bermekimab Concentration Over Time
Description: Serum bermekimab concentration over time were reported. Data are presented by individual dose of investigational medicinal product received by participants during active treatment period as preplanned in protocol.
Time Frame: Pre-dose at Week 0, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, and Week 36
Population: The pharmacokinetic (PK) analysis set included all participants who had received at least 1 dose of bermekimab and had at least 1 valid blood sample drawn for PK analysis. Here, "n (number analyzed)" specifies number of participants who were analyzed at the specified timepoint and '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per mililiters (mcg/mL)
Arm/Group | Placebo Then Bermekimab 700 mg | Bermekimab 350 mg | Bermekimab 700 mg Then Bermekimab 700 mg (Non-responders) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders)
Number analyzed (Participants) | 19 | 33 | 22 | 3 | 5
micrograms per mililiters (mcg/mL)
  Week 0: number analyzed (Participants) | 0 | 33 | 22 | 3 | 5
  Week 0 |  | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Week 1: number analyzed (Participants) | 0 | 32 | 22 | 2 | 4
  Week 1 |  | 24.80 (10.156) | 44.61 (16.945) | 36.88 (2.831) | 34.96 (11.796)
  Week 4: number analyzed (Participants) | 0 | 27 | 21 | 3 | 5
  Week 4 |  | 37.85 (19.347) | 75.65 (35.815) | 83.07 (46.927) | 71.15 (29.254)
  Week 8: number analyzed (Participants) | 0 | 24 | 21 | 3 | 5
  Week 8 |  | 42.33 (20.880) | 81.25 (41.734) | 80.72 (40.377) | 76.88 (32.047)
  Week 12: number analyzed (Participants) | 0 | 19 | 20 | 3 | 5
  Week 12 |  | 46.90 (19.759) | 81.17 (42.878) | 83.89 (21.875) | 74.06 (32.283)
  Week 16: number analyzed (Participants) | 18 | 18 | 21 | 3 | 5
  Week 16 | 0.00 (0.000) | 51.26 (19.349) | 80.56 (46.644) | 83.35 (43.518) | 77.95 (47.186)
  Week 20: number analyzed (Participants) | 14 | 14 | 18 | 3 | 4
  Week 20 | 86.49 (43.182) | 50.91 (20.004) | 79.51 (50.180) | 82.14 (21.151) | 38.73 (19.023)
  Week 24: number analyzed (Participants) | 12 | 11 | 12 | 3 | 4
  Week 24 | 90.40 (51.619) | 55.55 (24.609) | 65.57 (31.614) | 45.13 (31.291) | 23.93 (17.506)
  Week 28: number analyzed (Participants) | 6 | 7 | 9 | 2 | 2
  Week 28 | 99.41 (58.863) | 58.31 (24.150) | 62.20 (30.876) | 68.88 (13.172) | 2.02 (1.742)
  Week 32: number analyzed (Participants) | 2 | 7 | 2 | 1 | 1
  Week 32 | 30.13 (23.807) | 48.68 (21.937) | 12.95 (18.318) | 56.96 (NA) — NA indicates that standard deviation was not calculable because only one participant was involved in the analysis. | 38.84 (NA) — NA indicates that standard deviation was not calculable because only one participant was involved in the analysis.
  Week 36: number analyzed (Participants) | 0 | 6 | 2 | 1 | 0
  Week 36 |  | 7.31 (6.821) | 0.57 (0.813) | 4.44 (NA) — NA indicates that standard deviation was not calculable because only one participant was involved in the analysis. |

8. Secondary Outcome: Number of Participants With Anti-Bermekimab Antibodies
Description: Number of participants with anti-bermekimab antibodies were reported. Data are presented by individual dose of investigational medicinal product received by participants during active treatment period as preplanned in protocol.
Time Frame: Up to Week 36
Population: The immunogenicity analysis set included all participants who had received at least 1 dose of bermekimab and who had at least 1 sample obtained after their first dose of bermekimab for the detection of antibodies to bermekimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then Bermekimab 700 mg | Bermekimab 350 mg | Bermekimab 700 mg Then Bermekimab 700 mg (Non-responders) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders)
Number analyzed (Participants) | 19 | 33 | 22 | 3 | 5
Participants | 1 | 9 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 36 for serious and other (non-serious) adverse events; all-cause mortality: from screening up to end of study (up to Week 40)
Description: The safety analysis set included all participants who received at least 1 dose of study intervention.
Arm/Group | Placebo | Bermekimab 350 mg | Bermekimab 700 mg | Dupilumab | Placebo Then Bermekimab 700 mg | Bermekimab 350 mg Then Bermekimab 350 mg | Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) | Dupilumab Then Dupilumab 300 mg (Responders) | Dupilumab Then Bermekimab 700 mg (Non-Responders)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/67 | 0/65 | 0/19 | 0/21 | 0/22 | 0/3 | 0/5 | 0/27 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33 | 2/67 | 0/65 | 0/19 | 0/21 | 0/22 | 0/3 | 0/5 | 0/27 | 0/11
Other Adverse Events (participants affected / at risk) | 15/33 | 15/33 | 29/67 | 20/65 | 7/19 | 7/21 | 8/22 | 2/3 | 2/5 | 9/27 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Bermekimab 350 mg (N=33) | Bermekimab 700 mg (N=67) | Dupilumab (N=65) | Placebo Then Bermekimab 700 mg (N=19) | Bermekimab 350 mg Then Bermekimab 350 mg (N=21) | Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders) (N=22) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) (N=3) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) (N=5) | Dupilumab Then Dupilumab 300 mg (Responders) (N=27) | Dupilumab Then Bermekimab 700 mg (Non-Responders) (N=11)
Auricular Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Bermekimab 350 mg (N=33) | Bermekimab 700 mg (N=67) | Dupilumab (N=65) | Placebo Then Bermekimab 700 mg (N=19) | Bermekimab 350 mg Then Bermekimab 350 mg (N=21) | Bermekimab 700 mg Then Bermekimab 700 mg (Non-Responders) (N=22) | Bermekimab 700 mg Then Bermekimab 700 mg (Responders) (N=3) | Bermekimab 700 mg Then Bermekimab 350 mg (Responders) (N=5) | Dupilumab Then Dupilumab 300 mg (Responders) (N=27) | Dupilumab Then Bermekimab 700 mg (Non-Responders) (N=11)
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Erythema (General disorders) | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 4 | 2 | 1 | 2 | 5 | 3 | 3 | 1 | 1 | 1 | 2
Eczema Impetiginous (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lice Infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 8 | 6 | 1 | 0 | 3 | 0 | 0 | 4 | 2
Oral Herpes (Infections and infestations) | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pilonidal Cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 4 | 4 | 1 | 1 | 1 | 1 | 0 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 5 | 5 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 4 | 3 | 11 | 4 | 0 | 1 | 4 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT04791319/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT04791319/SAP_001.pdf